CLINICAL TRIAL: NCT06722001
Title: Comparing the Effectiveness of Brief Behavioral Treatment of Insomnia(BBTI) for Nursing Students and Nursing Staff Using Interactive E-books and Traditional Education Methods - a Randomized Clinical Trial
Brief Title: Comparing of Using Interactive E-books and Traditional Education Methods for Nursing Students and Nursing Staff
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Tsai-Wei Huang, professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: TMU_ebook
Record Dates: First submitted 2023-09-22; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Efficacy, Self; Satisfaction, Personal
Keywords: Brief Behavioral Treatment of Insomnia; e-book; Insomnia treatment
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional group (Active Comparator): The traditional group members will obtain traditional paper leaflets and oral health education.
  Interventions: Behavioral: traditional paper handout
- "Brief insomnia intervention" group (Experimental): The "Brief insomnia intervention" group will study the interactive e-book.
  Interventions: Behavioral: The "Brief insomnia intervention" interactive e-book

INTERVENTIONS:
Behavioral: The "Brief insomnia intervention" interactive e-book — The control group learned through paper health education leaflets and traditional oral explanations; the experimental group used interactive e-books to intervene in learning Brief Behavioral Treatment of Insomnia.
  Arms: "Brief insomnia intervention" group
Behavioral: traditional paper handout — The control group learned through paper health education leaflets and traditional oral explanations; the experimental group used interactive e-books to intervene in learning Brief Behavioral Treatment of Insomnia.
  Arms: Traditional group

SUMMARY:
Cancer-related comorbidities are a major focus of care for medical staff, especially the incidence of "insomnia" in cancer patients should not be underestimated, and the treatment of cancer-related insomnia by clinical medical staff is often limited to verbal instructions and suggestions, lacking routine and a systematic process. Although "Cognitive behavioral treatment for insomnia (CBTI)" is widely used, due to the limitation of personnel and high time cost, later generations improved "Brief Behavioral Treatment of Insomnia (BBTI)", which not only broadens the clinical application but also increases the patient's willingness to cooperate.

In recent years, the integration of technology into teaching has become a trend. Among them, interactive e-books are widely used. It not only enhances users' learning motivation and interest but also is effective in building practical confidence. It can also customize course content according to different needs.

The purpose of this study is to compare the effectiveness of using interactive e-book teaching and traditional teaching methods to learn Brief Behavioral Treatment of Insomnia. The object is aimed at nursing students and clinical nurses. An experimental research design is adopted. A total of 165~180 clinical nurses and university nursing students will be pre-selected and randomly assigned to the control group or the experimental group. The control group learned through paper health education leaflets and traditional oral explanations; the experimental group used interactive e-books to intervene in learning Brief Behavioral Treatment of Insomnia, the subjects needed to fill out the pre-test and post-test questionnaires before and after the experiment to compare the difference in the learning effects of the two groups of subjects, and expect that the group using interactive e-book will have better learning effects and course satisfaction.

DETAILED DESCRIPTION:
Cancer-related comorbidities are a major focus of care for medical staff, especially the incidence of "insomnia" in cancer patients should not be underestimated, and the treatment of cancer-related insomnia by clinical medical staff is often limited to verbal instructions and suggestions, lacking routine and a systematic process. Although "Cognitive behavioral treatment for insomnia (CBTI)" is widely used, due to the limitation of personnel and high time cost, later generations improved "Brief Behavioral Treatment of Insomnia (BBTI)", which not only broadens the clinical application but also increases the patient's willingness to cooperate.

In recent years, the integration of technology into teaching has become a trend. Among them, interactive e-books are widely used. It not only enhances users' learning motivation and interest but also is effective in building practical confidence. It can also customize course content according to different needs.

The purpose of this study is to compare the effectiveness of using interactive e-book teaching and traditional teaching methods to learn Brief Behavioral Treatment of Insomnia (BBTI). The object is aimed at nursing students and clinical nurses. An experimental research design is adopted. A total of 165~180 clinical nurses and university nursing students will be pre-selected and randomly assigned to the control group or the experimental group. The control group learned through paper health education leaflets and traditional oral explanations; the experimental group used interactive e-books to intervene in learning Brief Behavioral Treatment of Insomnia (BBTI), the subjects needed to fill out the pre-test and post-test questionnaires before and after the experiment to compare the difference in the learning effects of the two groups of subjects, and expect that the group using interactive e-book will have better learning effects and course satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Nursing students older than 20 years old.
2. Clinical nurses worked in the hospital more than three months.

Exclusion Criteria:

1. cognitive disabilities
2. incomplete behavioral ability

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Cognition knowledge scale | change in learning outcomes between baseline and 1 week
  learning Cognition knowledge outcomes from Brief Behavioral Treatment of Insomnia. higher score higher cognition knoeledge.
Confidence scale | change in learning outcomes between baseline and 1 week.
  learning Confidence outcomes from Brief Behavioral Treatment of Insomnia. higher score higher confidence.
Satisfied from learning | change in learning outcomes between baseline and 1 week.
  learning Satisfaction from Brief Behavioral Treatment of Insomnia. higher score higher satisfaction.

IPD SHARING:
Plan to Share IPD: No